CLINICAL TRIAL: NCT00189774
Title: Nateglinide: a Double Blind Add-on Study With Pioglitazone for Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Ajinomoto USA, INC. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 026-CL-004
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type II
Keywords: nateglinide; pioglitazone; combination drug therapy; treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Nateglinide

INTERVENTIONS:
Drug: nateglinide

SUMMARY:
The purpose of this study is to investigate the superiority of nateglinide over placebo for inadequately controlled type 2 diabetic patients with pioglitazone treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus under the treatment with pioglitazone

Exclusion Criteria:

* Patients who cannot follow the diet therapy and/or exercise therapy
* Type 1 diabetes mellitus

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Astellas Pharma Inc
Locations (7):
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Tohoku Region